CLINICAL TRIAL: NCT02939001
Title: Evaluating the Effect of Laser Vision Surgery, Phakic Intraocular Lens Implantation, Cataract Surgery, and Pupil Dilation on the Iris Recognition Scanner Function of Smartphone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-2016-0049
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Cataract; Myopia; Myopic Astigmatism
MeSH Terms: conditions — Cataract; Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ophthalmic surgery group (Experimental): Ophthalmic surgery group (refractive surgery, phakic Intraocular Lens implantation, and cataract surgery)
  Interventions: Device: iris recognition scanner

INTERVENTIONS:
Device: iris recognition scanner
  Other Names: Galaxy Note 7 (Smartphone)

SUMMARY:
This study included patients who visit for refractive surgery (photorefractive keratectomy, photorefractive keratectomy with with corneal collagen cross linking, laser in situ keratomileusis, small incision lenticule extraction), phakic Intraocular Lens implantation (Implantable Collamer Lens, artiflex), and cataract surgery. Patients will be examined whether iris recognition scanner of smartphone works before and after surgery. In addition, before and after pupil dilation (5mm, 6mm, 7mm, 8mm), patients will be examined whether iris recognition scanner of smartphone works well.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visit for refractive surgery (photorefractive keratectomy, photorefractive keratectomy with with corneal collagen cross linking, laser in situ keratomileusis, small incision lenticule extraction)
* phakic Intraocular Lens implantation (Implantable Collamer Lens, artiflex)
* cataract surgery.
* age of 20~90

Exclusion Criteria:

* history of previous ocular or intraocular surgery
* glaucoma or ocular hypertension, ocular infection, non-dry eye ocular inflammation, ocular allergy, autoimmune disease
* history of iris damage during ocular surgery or previous trauma
* wearing contact lenses during the study period
* presence of current punctal occlusion
* pregnancy, lactating women, and children

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
capability of iris recognition scanner | 1 day before the surgery
  Patients will be examined whether iris recognition scanner of smartphone works 1 day before refractive surgery (photorefractive keratectomy, photorefractive keratectomy with corneal collagen cross linking, laser in situ keratomileusis, small incision lenticule extraction), phakic Intraocular Lens implantation (Implantable Collamer Lens, artiflex), and cataract surgery.
capability of iris recognition scanner | 1 week after the surgery
  Patients will be examined whether iris recognition scanner of smartphone works 1 week after refractive surgery (photorefractive keratectomy, photorefractive keratectomy with corneal collagen cross linking, laser in situ keratomileusis, small incision lenticule extraction), phakic Intraocular Lens implantation (Implantable Collamer Lens, artiflex), and cataract surgery.

SECONDARY OUTCOMES:
pupil dilation | 1 day before pupil dilation
  Patients will be examined whether iris recognition scanner of smartphone works well 1 day before pupil dilation.
pupil dilation | 1 week after the surgery
  Patients will be examined whether iris recognition scanner of smartphone works well 1 week after before pupil dilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No